CLINICAL TRIAL: NCT03279744
Title: A Prospective, Single-Arm, Open-Label, Phase II. Study to Evaluate the Efficacy and Safety of Photodynamic Therapy Using Radion™-Pdt in Patients With Oral Precancerous Lesion (Oral Verrucous Hyperplasia or Oral Erythroleukoplakia)
Brief Title: A Study to Evaluate the Efficacy and Safety of Radion™-Pdt in Patients With Oral Precancerous Lesion
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pharma Power Biotec Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRC241001
Record Dates: First submitted 2017-09-08; First posted 2017-09-12 (Actual); Last update posted 2020-01-02 (Actual); Status verified 2019-12

CONDITIONS: Erythroleukoplakia of Mouth; Verrucous Hyperplasia of Oral Mucosa
Keywords: Oral Verrucous Hyperplasia; Oral Erythroleukoplakia

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single-Arm (Experimental): Radion™-pdt
  Interventions: Drug: Radion™-pdt

INTERVENTIONS:
Drug: Radion™-pdt — The Radion™-pdt will be applied topically to the lesion. The Radion™-pdt applied dosage is about 0.1 mL/cm^2 and properly cover the entire lesion.

SUMMARY:
A Prospective, Single-Arm, Open-Label, Phase II Study to Evaluate the Efficacy and Safety of Photodynamic Therapy Using Radion™-pdt in Patients with Oral Precancerous Lesion (Oral Verrucous Hyperplasia or Oral Erythroleukoplakia).

DETAILED DESCRIPTION:
This is a single-center, single-arm, open-label study to evaluate the efficacy and safety of topical Radion™-pdt for treatment of patients with oral verrucous hyperplasia (OVH) or oral erythroleukoplakia (OEL).

Total duration of the study will be up to 40 weeks (from screening throughout study until completion) as follows:

* Screening (within 2 weeks before dosing)
* Treatment period (up to 14 weeks)
* Safety follow-up period (within 2 weeks after final treatment)
* Follow-up period (final treatment plus 4 weeks, 8 weeks, 16 weeks and 24 weeks respectively) All enrolled patients will receive up to 8 treatments (once every two weeks) during a maximum of 14-week study treatment period. The treated lesion will be clinically evaluated and documented (clinical photograph) at each treatment visit.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged ≥20 years old;
2. Patient with oral verrucous hyperplasia (OVH) or oral erythroleukoplakia (OEL) lesions with histological evidence of oral precancerous lesions. Besides, patients should have at least one lesion whose size should not exceed 4 cm in the greatest diameter and the distance between two lesions should not less than 1 cm.
3. Patient who is willing and able to comply with study procedures and sign informed consent

Exclusion Criteria:

1. Patients with history of hypersensitivity to any photosensitizer (including 5-aminolevulinic acid HCl or porphyrins), acute or chronic types of porphyria;
2. Record of previous unsuccessful treatment with photodynamic therapy;
3. Patients who have been diagnosed as having oral cancer or carcinoma in situ;
4. Patients who have a history or evidence of a medical condition that would expose them to an undue risk of a significant adverse event during the course of the trial, including but not limited to hepatic, renal, respiratory, cardiovascular, endocrine, immune, neurological, hematological, gastrointestinal or psychiatric disease as determined by the clinical judgment of the investigator;
5. Patients with impaired hepatic function (defined as AST and/or ALT > 2× the upper limit of normal values), and/or impaired renal function (defined as serum creatinine > 1.5 mg/dL);
6. Female patient of childbearing potential who:

   * is lactating; or
   * has positive urine pregnancy test at visit -1; or
   * refuses to adopt reliable method of contraception during the study;
7. Patient has received any other investigational agent within 28 days or 5 half-lives, whichever is longer, prior to the first photodynamic therapy;
8. Patient has a history of illegal substance abuse, drug addiction or alcoholism within 24 weeks prior to the study.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2017-09-06 (Actual); Primary Completion 2019-09-04 (Actual); Study Completion 2019-12-20 (Actual)

PRIMARY OUTCOMES:
The primary efficacy endpoints: the complete response rate is higher or equal to 70% of total | 2-week safety follow-up period after last treatment
  The complete response rate at the end of treatment will be calculated by the proportion of complete response patients in total. The primary efficacy endpoints will be summarized by examining whether the complete response rate is higher or equal to 70% of total.
  Complete response (CR): lack of detectable lesion confirmed by visual evaluation.

CONTACTS AND LOCATIONS:
Overall Officials: Hsin-Ming Chen, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Zhongzheng Dist, Taiwan